CLINICAL TRIAL: NCT05392738
Title: Visual Function and Patient Satisfaction in Glaucoma or Ocular Hypertensive Patients Undergoing Simultaneous Cataract Surgery and i-Stent Implantation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Clínica Rementería (Other)
Responsible Party: Sponsor
Other Study IDs: 22/265-O_P
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Lenses, Intraocular; Glaucoma Filtration Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Vivity with i-Stent: Patients with Glaucoma or Ocular Hypertension undergoing simultaneous cataract and i-Stent implantation, with Vivity intraocular lens
  Interventions: Device: I-Stent implantation
- Glaucoma with Vivity: Patients with Glaucoma or Ocular Hypertension undergoing isolated phacoemulsification with Vivity intraocular lens
- Healthy with Vivity: Patients with undergoing isolated phacoemulsification with Vivity intraocular lens

INTERVENTIONS:
Device: I-Stent implantation — I-Stent implantation
  Groups: Vivity with i-Stent

SUMMARY:
New extended depth of focus intraocular lenses (IOLs) are being used in a broader spectrum of patients than trifocal IOLs. The purpose of this study is to evaluate visual improvement after cataract surgery in patients with glaucoma or ocular hypertension undergoing simultaneous cataract surgery with i-Stent implantation with the implantation of a Vivity IOL. Results will be compared with a group of glaucoma or ocular hypertension undergoing isolated cataract surgery with Vivity implantation, as well as with patients with no pathology undergoing cataract surgery and Vivity implantation

DETAILED DESCRIPTION:
The purpose of this study is to report in detail visual function and patient satisfaction, as well as the need for spectacle correction, in patients with glaucoma and ocular hypertension undergoing cataract surgery with bilateral implantation of an extended depth of focus IOL, the Vivity IOL. The study also seeks to determine if there are differences in the speed of visual improvement between patients undergoing isolated cataract surgery and patients undergoing simultaneous i-Stent implantation. Results will also be compared with a group of patients with no ocular pathology undergoing cataract surgery with Vivity implantation.

Patients will be asked to join the study once the type of surgery (isolated phacoemulsification versus phacoemulsification combined with i-Stent implantation) and the type of lens to be implanted (monofocal, EDoF, trifocal) has been agreed between ophthalmologist and patient. Therefore, inclusion in the study will have no influence on surgical indication.

Once informed consent has been signed, the patient will be included in the study.

Explorations specific for the study will be performed 3 and 12 months after surgery and include:

Defocus curves Contrast sensitivity Self-reported photic phenomena Need for spectacle correction Satisfaction measured with the Catquest SF9 questionnaire

Besides study-specific procedures, the following explorations which are standard of care will be performed one day, one week and one month after surgery:

Uncorrected binocular visual acuity for distance, intermediate and near distances Monocular distance corrected and uncorrected visual acuity Residual subjective refraction Slit-lamp examination Intraocular pressure and number of hypotensive drugs required Description of any intra- or postsurgical complications

ELIGIBILITY:
Inclusion Criteria: Bilateral cataract surgery with Vivity implantation with or without i_STent implantation

Exclusion Criteria: Ocular disease other than glaucoma

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with glaucoma or ocular hypertension or healthy subjects undergoing bilateral cataract surgery with Vivity intraocular lens implantation with or without i-Stent implantation
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Binocular uncorrected distance visual acuity | Three months after surgery
  Binocular uncorrected distance visual acuity
Binocular uncorrected intermediate visual acuity | Three months after surgery
  Binocular uncorrected intermediate visual acuity
Binocular uncorrected near visual acuity | Three months after surgery
  Binocular uncorrected near visual acuity

SECONDARY OUTCOMES:
Binocular uncorrected distance visual acuity | One month after surgery
  Binocular uncorrected distance visual acuity
Binocular uncorrected intermediate visual acuity | One month after surgery
  Binocular uncorrected intermediate visual acuity
Binocular uncorrected near visual acuity | One month after surgery
  Binocular uncorrected near visual acuity
Contrast sensitivity | Three months after surgery
  Contrast sensitivity
Need for spectacle correction | Three months after surgery
  Need for spectacle correction
Patient satisfaction | Three months after surgery
  Patient satisfaction evaluated with the Catquest SF9 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Puerto, MD, Principal Investigator — Clínica Rementería
Locations (1):
- Clínica Rementería, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided